CLINICAL TRIAL: NCT04471974
Title: A Phase 2 Study of BET Bromodomain Inhibitor ZEN-3694 in Combination With Enzalutamide Plus Pembrolizumab in Metastatic Castration Resistant Prostate Cancer
Brief Title: ZEN-3694, Enzalutamide, and Pembrolizumab for the Treatment of Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rahul Aggarwal (Other)
Collaborators: Zenith Epigenetics (Industry); Merck Sharp & Dohme LLC (Industry); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Rahul Aggarwal, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20551; NCI-2020-04495 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Adenocarcinoma; Metastatic Prostate Small Cell Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Safety Cohort (Experimental): Patients receive 96mg pembrolizumab IV over 30 minutes on day 1, BET bromodomain inhibitor ZEN-3694 PO QD and enzalutamide PO QD on days 1-21. Patients not on enzalutamide prior to study enrollment or have previously discontinued enzalutamide receive BET bromodomain inhibitor ZEN-3694 beginning on day 1 of cycle 2. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Drug: Enzalutamide; Biological: Pembrolizumab
- Cohort A: Transdifferentiated mCRPC (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1, BET bromodomain inhibitor ZEN-3694 PO QD and enzalutamide PO QD on days 1-21. Patients not on enzalutamide prior to study enrollment or have previously discontinued enzalutamide receive BET bromodomain inhibitor ZEN-3694 beginning on day 1 of cycle 2. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Drug: Enzalutamide; Biological: Pembrolizumab
- Cohort B: mCRPC without evidence of transdifferentiation (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1, BET bromodomain inhibitor ZEN-3694 PO QD and enzalutamide PO QD on days 1-21. Patients not on enzalutamide prior to study enrollment or have previously discontinued enzalutamide receive BET bromodomain inhibitor ZEN-3694 beginning on day 1 of cycle 2. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Drug: Enzalutamide; Biological: Pembrolizumab

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial investigates how well ZEN-3694, enzalutamide, and pembrolizumab work in treating patients with castration-resistant prostate cancer that has spread to other places in the body (metastatic). ZEN-3694 blocks the expression of the MYC gene to prevent cellular growth in certain types of tumors, including castrate resistant prostate cancer. Enzalutamide has been shown to block testosterone from reaching prostate cancer cells by binding to a receptor on prostate cancer cells, called androgen receptors. This works similar to a lock and key. When enzalutamide (key) inserts into the androgen receptor (lock) testosterone cannot attach to the androgen receptor, which slows the growth of tumor cells and may cause them to shrink. Pembrolizumab is a monoclonal antibody (proteins that can protect the body from foreign organisms, such as bacteria and viruses) designed to block a specific control switch which may be activated by tumor cells to overcome the body's natural immune system defenses. It also enhances the activity of the body's immune cells against tumor cells. The purpose of this study is to find out the effects ZEN-3694, enzalutamide, and pembrolizumab on patients with metastatic castration-resistant prostate cancer who have previously experienced disease progression.

DETAILED DESCRIPTION:
Patients with metastatic castration resistant prostate cancer (mCRPC) who had prior disease progression on at least one second generation androgen signaling inhibitor, including abiraterone, apalutamide, darolutamide, and/or enzalutamide and have clinicogenomic evidence of transdifferentiated mCRPC (Cohort A) or mCRPC without transdifferentiation (Cohort B). Prior to enrollment in Phase 2 (Cohort A and B), a safety lead-in cohort of 6 patients with metastatic CRPC will be enrolled. Accrual will proceed to Phase 2 if < 33% of patients (0/6 or 1/6 patients) experiences a dose-limiting toxicity during Cycle 1.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1, BET bromodomain inhibitor ZEN-3694 orally (PO) once daily (QD) and enzalutamide PO QD on days 1-21. Patients not on enzalutamide prior to study enrollment or have previously discontinued enzalutamide receive BET bromodomain inhibitor ZEN-3694 beginning on day 1 of cycle 2. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 90 days until death or study completion or loss to follow-up, whichever occurs first.

PRIMARY OBJECTIVE:

I. To determine the composite response rate in Cohort A and Cohort B study population.

SECONDARY OBJECTIVES:

I. To determine the objective response rate and median duration of response in each study cohort.

II. To determine the median progression free survival and 6-month progression-free survival rate.

III. To determine the prostate-specific antigen (PSA) 50 (PSA50) response proportion in each study cohort.

IV. To determine the median overall survival of each cohort. V. To determine the safety of the treatment combination.

EXPLORATORY OBJECTIVES:

I. To explore the association between baseline metastatic tumor characteristics including treatment-emergent small cell neuroendocrine carcinoma (t-SCNC), androgen receptor (AR), retinoblastoma tumor suppressor gene (RB1) loss, and immune response transcriptional signatures with clinical outcomes.

II. To evaluate modulation of AR transcriptional activity, expression of t-SCNC markers, and immune parameters including tumor-infiltrating lymphocytes and PD-L1 expression in evaluable paired tumor biopsies.

III. To evaluate the association between baseline and change from baseline in peripheral blood biomarkers including T cell subsets, T cell repertoire, and inhibitors of bromodomain extraterminal protein (BETi) whole blood ribonucleic acid (RNA) panel with clinical outcomes.

IV. To evaluate the association between baseline or change from baseline in gallium Ga 68 citrate (68Ga-citrate) positron emission tomography (PET) with subsequent clinical outcomes.

V. To compare efficacy outcomes (composite response, PSA50 response, objective response, progression-free survival (PFS), and overall survival (OS)) between cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed prostate adenocarcinoma at the time of diagnosis, with subsequent development of metastatic castration-resistant prostate cancer. Patients with de novo small cell prostate cancer at the time of diagnosis are excluded from study participation
2. Evidence of disease progression by PSA and/or radiographic progression by Prostate Cancer Working Group 3 (PCWG3) criteria at the time of study entry
3. Patients must be evaluable for the primary endpoint of composite response, and must have either serum PSA > 2 ng/mL during Screening and/or measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
4. Safety lead-in only:

   1. Metastatic castration resistant prostate cancer with evidence of disease progression by PCWG3 criteria at study entry
   2. Progression on at least one prior androgen signaling inhibitor (e.g. abiraterone/prednisone, enzalutamide, apalutamide, darolutamide)
   3. No prior chemotherapy for the treatment of metastatic castration-resistant prostate cancer (mCRPC). Prior chemotherapy administered in the castration-sensitive setting is allowed provided last dose of chemotherapy is > 6 months prior to cycle 1 day 1 (C1D1)
5. Phase 2 Cohort A (transdifferentiated mCRPC) only:

   a. Participants must have clinicogenomic evidence of treatment emergent small cell neuroendocrine prostate cancer as defined by one or more of the following.

   i. Histologic evidence of small cell neuroendocrine prostate cancer on metastatic tumor biopsy and/or

   ii. Presence of loss-of-function mutation or deletion of RB1 on a Clinical Laboratory Improvement Act (CLIA)-approved genomic-sequencing platform and/or

   iii. Low PSA secretors as defined by meeting all of the following criteria during screening period -
   * Serum PSA >=2 ng/mL,
   * Radiographic progression by PCWG3 criteria,
   * Presence of > 5 metastases on conventional imaging and/or

   iv. Presence of at least one soft tissue lesion measuring > 1 cm that is negative on PSMA PET. A negative lesion on PSMA PET is defined as uptake below the background uptake in the liver.

   b. No more than two prior lines of chemotherapy administered in the mCRPC setting. Chemotherapy administered in the castration-sensitive setting does not count towards this limit.

   c. Measurable disease by RECIST 1.1 criteria.
6. Phase 2 Cohort B (mCRPC without transdifferentiation) only:

   1. Patients must not meet any criteria of transdifferentiation as outlined above
   2. Progression on at least one prior androgen signaling inhibitor (e.g. abiraterone/prednisone, enzalutamide, apalutamide, darolutamide)
   3. No prior chemotherapy for the treatment of mCRPC. Prior chemotherapy administered in the castration-sensitive setting is allowed provided last dose of chemotherapy is > 6 months prior to C1D1
7. Castrate level of serum testosterone at study entry (< 50 ng/dL). Patients without prior bilateral orchiectomy are required to remain on luteinizing hormone-releasing hormone (LHRH) analogue treatment for duration of study
8. No other systemic anti-cancer therapies administered other than LHRH analogue within 14 days or, 5 half-lives, whichever is shorter, prior to initiation of study treatment. Adverse events related to prior anti-cancer treatment must have recovered to grade =< 1 with the exception of any grade alopecia and grade =< 2 neuropathy

   a. Patients receiving enzalutamide prior to study entry may continue treatment at their current enzalutamide dose level without requirement for wash-out period
9. Age >= 18 years
10. Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky performance status >= 70%)
11. Demonstrates adequate organ function as defined below:

    * Absolute neutrophil count >= 1,500/ per microliter (mcL)
    * Platelets >= 100,000/mcL
    * Hemoglobin >= 9.0 g/dL
    * Total bilirubin =< 1.5 x institutional upper limit of normal, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits
    * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT) =< 3 x institutional upper limit of normal (=< 5 x upper limit of normal (ULN) in presence of liver metastases)
    * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 3 x institutional upper limit of normal (=< 5 x ULN in presence of liver metastases)
    * Serum creatinine =< 1.5 x institutional upper limit of normal OR calculated creatinine clearance glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 , calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
12. Ability to understand a written informed consent document, and the willingness to sign it
13. Patients must agree to use adequate contraception prior to the study, for the duration of study participation, and 60 days after last administration of study treatment. Adequate contraception includes:

    1. Patients who are sexually active should consider their female partner to be of childbearing potential if she has experienced menarche and is not postmenopausal (defined as amenorrhea > 24 consecutive months) or has not undergone successful surgical sterilization. Even women who use contraceptive hormones (oral, implanted, or injected), an intrauterine device, or barrier methods (diaphragms, condoms, spermicide) should be considered to be of childbearing potential
    2. Patients who have undergone vasectomy themselves should also be considered to be of childbearing potential
    3. Acceptable methods of contraception include continuous total abstinence, or double-barrier method of birth control (e.g. condoms used with spermicide, or condoms used with oral contraceptives). Periodic abstinence and withdrawal are not acceptable methods of contraception
14. Patients must be willing to undergo metastatic tumor biopsy during screening. If no metastatic lesion is safely accessible to tumor biopsy, this requirement will be waived. Bone or soft tissue lesion is allowed, but soft tissue will be prioritized. If a patient has archival tissue obtained within 90 days of C1D1 the requirement for fresh tumor biopsy will be waived

Exclusion Criteria:

1. Has participated in a study of an investigational product and received study treatment or used an investigational device other than those specified in the protocol within 2 weeks of C1D1
2. Hypersensitivity to ZEN-3694, pembrolizumab, enzalutamide, or any of its excipients
3. Has received prior radiotherapy within 2 weeks of C1D1. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
4. Receipt of prior pembrolizumab or another immune checkpoint inhibitor (e.g. nivolumab, ipilimumab). Prior treatment with sipuleucel-T is allowed
5. Receipt of a radiopharmaceutical (e.g. radium-223, 177Lu-prostate-specific membrane antigen (PSMA) within 6 weeks prior to C1D1
6. Prior treatment with a bromodomain inhibitor (BETi)
7. Individuals with concurrent second malignancy requiring active treatment at study entry. Non-melanoma skin cancer, non-muscle invasive bladder cancer, and other carcinomas-in-situ are allowable exceptions
8. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients on low dose oral weekly methotrexate are allowed. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) or treatment with drugs (e.g. methimazole, neomercazol, carbamazole, etc.) that function to decrease the generation of thyroid hormone by a hyper-functioning thyroid gland (e.g., in Graves' disease) is not considered a form of systemic treatment of an autoimmune disease
9. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
10. Cardiac condition as defined as one or more of the following:

    1. QT interval by Fridericia (QTcF) > 480 ms (machine or manual read allowed)
    2. Uncontrolled supraventricular arrhythmia or ventricular arrhythmia requiring treatment
    3. New York Heart Association (NYHA) congestive heart failure class III or IV
    4. History of unstable angina, myocardial infarction, or cerebrovascular accident within 6 months prior to C1D1
11. History of seizure or pre-disposing condition (e.g. brain metastases)
12. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy at a prednisone equivalent dose of > 10 mg daily or other form of immunosuppressive therapy within 7 days prior to first dose of study drug
13. Human immunodeficiency virus (HIV)-infected individuals on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial (screening not required in the absence of risk factors)
14. For participants with evidence of chronic hepatitis B virus (HBV) infection (positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb)), the HBV viral load must be undetectable at the time of study enrollment (screening not required in the absence of risk factors)
15. Chronic active hepatitis C virus (HCV) infection defined as positive viral load (screening not required in the absence of risk factors)
16. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/ interstitial lung disease
17. Has an active infection requiring intravenous antibiotics within 7 days prior to C1D1
18. Use of a prohibited concomitant medication within 7 days of C1D1
19. Major surgery within 28 days prior to C1D1. Minor procedures including biopsies, dental surgery, cataract surgery, or outpatient procedure are allowed
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite Response Rate | Up to 3 years
  Defined as either objective response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria (complete response (CR), partial response (PR)) or confirmed >= 50% decline from serum prostate-specific antigen (PSA) at baseline confirmed by repeat measurement performed ≥ 4 weeks later for each study cohort. To be considered evaluable for PSA50 response, patients must have a serum PSA >=2 ng/mL at baseline. To be considered evaluable for objective response, patients must have measurable soft tissue disease by RECIST 1.1 criteria on baseline scan assessment. The composite response rate along with 95% confidence interval will be reported for participants in each study cohort.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years
  Objective response is defined as a complete response (CR), partial response (PR)) for the subset of patients with measurable soft tissue disease by RECIST 1.1 criteria. ORR will be reported along with 95% confidence interval for each study cohort. To be considered evaluable for objective response, patients must have measurable soft tissue disease by RECIST 1.1 criteria on baseline scan assessment Only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Median Duration of Response | Up to 3 years
  The duration of overall response is measured from the time measurement criteria are met for CR, PR, or stable disease (SD) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented. Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started. The median duration of response will be reported along with 95% confidence interval for each study cohort, for the subset of patients with measurable soft tissue disease by RECIST 1.1 criteria.
Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Will be determined for each cohort using Kaplan-Meier product limit method.
PSA50 response proportion | Up to 3 years
  PSA50 response is a >= 50% decline from baseline in serum PSA, confirmed by repeat measurement >= 4 weeks later. The PSA50 response proportion will be reported along with 95% confidence interval for each study cohort, for the subset of PSA-evaluable patients (serum PSA >= 2 ng/mL at baseline).
Overall survival (OS) | Up to 3 years
  The median overall survival along with 95% confidence interval will be determined from the date of first dose of protocol-defined therapy until death from any cause, using the Kaplan-Meier product limit method. Patients who withdraw from study will be censored for analysis of overall survival using the date of study withdrawal.
Incidence of treatment-related adverse events | Up to 30 days post-last dose
  All participants will be evaluable for toxicity from the time of their first protocol-defined treatment on C1D1. Will be recorded and severity graded using Common Terminology Criteria for Adverse Events version 5.0.The frequency and severity of adverse events will be descriptively reported

CONTACTS AND LOCATIONS:
Overall Officials: Rahul R Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - University of Chicago, Evergreen Park, Illinois
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No